CLINICAL TRIAL: NCT04554329
Title: Efficacy of Bandage Contact Lenses Versus Eye Patching in Early Postoperative Period of Müller's Muscle-conjunctival Resection
Brief Title: Bandage Contact Lenses Versus Eye Patching of Müller's Muscle-conjunctival Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Serhat Mangan, Medical Doctor, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HNEAH-KAEK 2019/116
Record Dates: First submitted 2020-08-07; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Eyelid Diseases
Keywords: patient comfort
MeSH Terms: conditions — Eyelid Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bandage contact lens (Active Comparator): A bandage contact lens was applied on the eye at the end of the surgery, and the eye was not covered with a patch.
  Interventions: Procedure: bandage contact lens
- eye patching (Active Comparator): Antibiotic eye ointment was applied on the eye, and the eye was covered with a patch at the end of the surgery.
  Interventions: Procedure: bandage contact lens

INTERVENTIONS:
Procedure: bandage contact lens — bandage contact lens

SUMMARY:
Patients with blepharoptosis who are treated with Müller's muscle-conjunctival resection (MMCR) may experience postoperative pain and discomfort related to the suture material on the palpebral conjunctiva. This study aims to compare the postoperative subjective complaints, such as pain and discomfort, with a visual analog scale (VAS) and objectively evaluate the cornea with a tear break-up time (TBUT) test and fluorescein staining following MMCR that was managed by either a bandage contact lens (BCL) or eye patching.

DETAILED DESCRIPTION:
Patients with blepharoptosis who are treated with Müller's muscle-conjunctival resection (MMCR) may experience postoperative pain and discomfort related to the suture material on the palpebral conjunctiva. This study aims to compare the postoperative subjective complaints, such as pain and discomfort, with a visual analog scale (VAS) and objectively evaluate the cornea with a tear break-up time (TBUT) test and fluorescein staining following MMCR that was managed by either a bandage contact lens (BCL) or eye patching.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had unilateral ptosis and underwent unilateral MMCR

Exclusion Criteria:

* Patients were excluded if they had previous eyelid surgery or had another known eye disease, such as ocular surface disorders, dry eye syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
patient comfort | 1 week
  VAS scores, (0: lowest; 10: highest)
patient comfort | 1 week
  TBUT score, (the minimum score was 0, and the maximum score was 15)

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpasa Numune Education and Research Hospital, Istanbul, Marmara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided